CLINICAL TRIAL: NCT05568342
Title: The Effect of Roy Adaptation-Based Nursing Intervention on Stress, Psychosocial Adjustment and Self-Care Power in Hemodialysis Patients: A Randomized Controlled Experimental Study
Brief Title: The Effect of Roy Adaptation-Based Nursing Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gaziantep Islam Science and Technology University (Other)
Responsible Party: Principal Investigator, Emine Karacan, Lecturer, Gaziantep Islam Science and Technology University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: Roy Adaptation Model
Record Dates: First submitted 2022-09-28; First posted 2022-10-05 (Actual); Last update posted 2022-10-05 (Actual); Status verified 2022-09

CONDITIONS: Hemodialysis Complication; Stress Disorders, Post-Traumatic; Psychosocial Impairment; Self Neglect
Keywords: Hemodialysis, Roy Adaptation Model, Stress, Self-Care Power, Psychosocial Adjustment
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Roy Group (Experimental): The population of the research consisted of 80 patients receiving outpatient dialysis treatment in the hemodialysis unit of a university hospital. In the sample of the study, those patients who came to the dialysis session on Monday-Wednesday-Friday were randomly assigned to the Roy group (experimental) (40 patients).
  Pre-test was applied to the patients in Roy and clinical groups using data collection tools. After the pre-test, the patients in the Roy group were trained 6 times in 3 months, twice a month, at home and in the clinic. Nursing interventions were performed using the Roy Adaptation Model in the trainings. At the end of the third month, the post-test data of both groups were collected. During the study, no training or intervention was given to the patients in the clinical group. The nursing education and interventions of this group were carried out by nurses working in the dialysis clinic within the scope of routine practices.
  Interventions: Behavioral: The Effect of Roy Adaptation-Based Nursing Intervention on Stress, Psychosocial Adjustment and Self-Care Power in Hemodialysis Patients: A Randomized Controlled Experimental Study
- Clinic Group (No Intervention): The population of the research consisted of 80 patients receiving outpatient dialysis treatment in the hemodialysis unit of a university hospital. In the sample of the study, those patients who came to the dialysis session on Tuesday-Thursday-Saturday were included in the Clinical group (control) (40 patients).
  Pre-test was applied to the patients in Roy and clinical groups using data collection tools. After the pre-test, the patients in the Roy group were trained 6 times in 3 months, twice a month, at home and in the clinic. Nursing interventions were performed using the Roy Adaptation Model in the trainings. At the end of the third month, the post-test data of both groups were collected. During the study, no training or intervention was given to the patients in the clinical group. The nursing education and interventions of this group were carried out by nurses working in the dialysis clinic within the scope of routine practices.

INTERVENTIONS:
Behavioral: The Effect of Roy Adaptation-Based Nursing Intervention on Stress, Psychosocial Adjustment and Self-Care Power in Hemodialysis Patients: A Randomized Controlled Experimental Study — Pre-test was applied to the patients in Roy and clinical groups using data collection tools. After the pre-test, the patients in the Roy group were trained 6 times in 3 months, twice a month, at home and in the clinic. Nursing interventions were performed using the Roy Adaptation Model in the trainings. At the end of the third month, the post-test data of both groups were collected. During the study, no training or intervention was given to the patients in the clinical group. The nursing education and interventions of this group were carried out by nurses working in the dialysis clinic within the scope of routine practices.
  Arms: Roy Group

SUMMARY:
Abstract Objective: The research was conducted to determine the effect of the nursing intervention, which was given to patients according to the Roy Adaptation Model, on patients' stress, psychosocial adjustment, and self-care power.

Methods: The population of the study, which was conducted as a randomized controlled experimental study, consisted of 80 patients receiving outpatient dialysis treatment in the hemodialysis unit of a university hospital. The patients from the population were included in the sample of the study in a randomized manner. The data were collected using the Descriptive Characteristics Form, the Hemodialysis Stressor Scale, the Self-Care Scale, and the Psychosocial Adjustment to Illness Scale.

Results: When the pre-tests between the groups were compared, hygienic self-care power, healthcare orientation, vocational environment, domestic environment, sexual relationships, extended family relations, social environment and total psychosocial adjustment levels changed significantly (p<0.05). When the post-tests were compared between the groups, no significant difference was found only in the mean of the mental state sub-dimension (p>0.05).

Conclusion: Interventions made according to the Roy Adaptation Model reduced the stress level of the patients, and increased their self-care power and psychosocial adjustment.

Keywords: Hemodialysis, Roy Adaptation Model, Stress, Self-Care Power, Psychosocial Adjustment

DETAILED DESCRIPTION:
1. Introduction and Objective Chronic Renal Failure (CKD) is a chronic and progressive deterioration in the functions of the kidney (Ammirati, 2020). Dialysis and renal transplantation applications play an important role in the treatment of CKD (Zhang and et al. 2020). However, dialysis is the most preferred treatment method because renal transplantation is not suitable for every patient and the risk of rejection is high (Imtiaz and Alam, 2021; Bleyer, 2022). Hemodialysis treatment is used in 70% of the patients in the world (Bello and et al. 2022) and in 76.9% of the patients in Turkey (Süleymanlar, 2020).

   While hemodialysis treatment saves patients from death and enables them to continue living, it also brings with it some physical, psychological, social and economic problems (Aksoy and Oğur, 2015). Loss of physical strength and endurance, body image disorder, fear of death, financial difficulties, diet, fluid intake, restricted activities, being dependent on machinery and hospital at certain days and hours of the week, invasive procedures applied in each session, loss of social relations, and dependence on medical treatment cause this disease to be perceived as an extreme source of stress, and changes caused by the disease in family and marital life increase the severity of the stress (Topbaş & Bingöl, 2017).

   The stress experienced negatively affects the psycho-social adaptation and self-care power of patients (Varol & Sivrikaya, 2018). While patients' non-compliance with treatment increases morbidity, mortality and economic problems (Sultan et al., 2022), inadequacy in self-care power causes problems in controlling the disease process and symptoms and meeting patients' own needs (Avanji et al., 2021; Gamze and Entertainment, 2013). Therefore, holistic nursing care has an important place in increasing the psycho-social adjustment and self-care power of hemodialysis patients.

   The use of models will guide nurses in providing standardization in holistic nursing care (Jasemi et al., 2017). The Roy Adaptation Model (RAM), one of the models widely used in nursing, creates a framework for determining the adaptation needs of individuals, families and groups, and focuses on the changes that occur in the adaptive system of the human and the environment. In this model, which includes four areas of adaptation: physiological, self-concept, role function and interdependence, the human being is defined as a biopsychosocial entity who is in constant interaction with his/her environment and is affected by stimuli (Roy et al., 2009). Associating the Roy Adaptation Model with patients undergoing hemodialysis treatment and providing training in line with this model may yield correct results in terms of nursing practice (Vicdan & Karabacak, 2014). In the literature, in the care of epilepsy (Erdoğan, 2021), cancer (Pehlivan et al., 2022), Covid-19 (Çaylar and Terzi, 2021), bariatric surgery (Guven et al., 2021) and many other diseases (Dağcan et al., 2021; Başayar et al., 2020; Yoldaş et al., 2019; Ilkaz et al., 2018), the Roy adaptation model was used. As a result of these studies, it was determined that patients' compliance with treatment increased and that nursing interventions gave positive results.

   In the literature, there are descriptive (Vicdan and Karabacak, 2014) and experimental studies (Vicdan and Karabacak, 2016) and case reports (Özdemir, 2022) studies showing the benefits of using the Roy adaptation model in hemodialysis patient education in terms of adaptation to illness. However, there is no experimental study evaluating stress, self-care power and psychosocial adaptation in hemodialysis patients by performing interventions according to the Roy adaptation model. For this reason, this study is important in terms of enabling patients to cope with stress and increasing their self-care power by increasing the adaptation to illness with the nursing interventions applied to the patients according to the Roy adaptation model.

   Objective The research was carried out to determine the effect of the nursing intervention given to patients according to the Roy Adaptation Model on patients' stress, psychosocial adjustment and self-care power and to contribute to patients and nursing interventions.

   The hypotheses in the post-test of the Roy group, which was applied according to the Roy adaptation model, are as follows:

   H1: Stress level is lower than the clinical group. H2: Self-care power level is higher than the clinical group. H3: Psychosocial adjustment level is higher than the clinical group.
2. Materials and Methods Location of the Research The study was conducted between 1 September and 30 November in the hemodialysis unit of a university hospital and at patients' homes.

2.1. Type of the Research The research was performed as a randomized controlled experimental study. Population and Sample of the Research The population of the research consisted of 80 patients receiving outpatient dialysis treatment in the hemodialysis unit of a university hospital. In the sample of the study, those patients who came to the dialysis session on Monday-Wednesday-Friday were randomly assigned to the Roy group (experimental) (40 patients), and those who came to the dialysis session on Tuesday-Thursday-Saturday were included in the Clinical group (control) (40 patients). The criteria for inclusion in the study were as follows: the absence of hearing and visual impairments that would prevent communication; no diagnosed psychiatric disorder; literacy; and Turkish proficiency.

2.1. Data Collection Tools 2.1.1. Descriptive Characteristics Form This form, prepared by the researchers, was created under the headings of socio-demographic characteristics (7 questions) and characteristics related to the disease (13 questions).

2.1.2. Hemodialysis Stressor Scale The scale developed by Baldree et al. (1982) was adapted to Turkish society by Kara (2006). The perceived physiological (6 items) and psychosocial stressors (23 items) associated with the treatment of hemodialysis patients are listed in the scale. The 5-point Likert scale is coded as "Always" (5 points), "Often" (4 points), "Sometimes" (3 points), "Rarely" (2 points), "Never" (1 points). The Physiological Hemodialysis Stressor sub-dimension score is between 6-30 points, the Psychosocial Hemodialysis Stressor sub-dimension score is between 23-115 points, and the total scale score is between 29-145. An increase in the score obtained from the scale indicates an increase in the perceived stress level. The total Cronbach alpha value of the scale is 0.77 (Kara,2006). The Cronbach's alpha value of our study was 0.85 in the pre-test group and 0.80 in the post-test group.

2.1.3. Self-Care Power Scale It is a scale developed by Ören (2010) for hemodialysis and peritoneal dialysis patients. The scale is a 3-point Likert-type scale consisting of 22 items and is scored between 0-2. The items 12, 22, 23, and 25 on the scale are reversed. Each item is answered as 'I always apply' (2 points), 'I sometimes apply' (1 point) and 'I do not apply at all' (0 points). The total score obtained from the scale is between 0-44. The scale has 5 sub-dimensions: Drug Use: 1,2,3,4,5,20, Diet: 8,9,10,11,12, Self-Monitoring: 6,7,13,14, Hygienic Care: 16,17 ,18,21, and Mental State 22,23,25. Scoring for the sub-dimensions is obtained by summing the item scores under each sub-dimension. At this point, drug use scores change between 0-12, diet scores change between 0-10, self-monitoring scores change between 0-8, hygienic care scores change between 0-4, and mental state scores change between 0-6. Low scores obtained as a result of the analysis indicate that self-care power is not good, whereas high scores indicate good self-care power. The Cronbach's alpha value of the whole scale was 0.75 in the hemodialysis group (Ören, 2014). The Cronbach's alpha value of our study was 0.70 in the pre-test group and 0.73 in the post-test group.

2.1.4. Psychosocial Adjustment to Illness-Self-Report Scale This scale, which was developed by Derogatis (1986) and evaluates psychosocial adjustment to illness, measures the interaction of individuals with other individuals and institutions that make up the socio-cultural environment. This scale, which was validated in Turkey by Adaylar (1995), consists of 46 items and 7 sub-dimensions. These sub-dimensions are Healthcare orientation, Vocational environment, Domestic environment, Sexual relationships, Extended Family Relations, Social Environment and Psychological distress. Each item is scored between 0-3. Major negative changes since illness are scored with 3 points, whereas no change or positive changes are scored with 0 points. The total score obtained from the scale is between 0-138. A low score on this scale indicates "good psychosocial adjustment" to illness, and a high score indicates "poor psychosocial adjustment" to illness. The Cronbach's alpha value of the whole scale was determined as 0.94 (Adaylar, 1995). The Cronbach's alpha value of our study was 0.91 in the pre-test group and 0.94 in the post-test group.

2.2. Data Collection Method Pre-test was applied to the patients in Roy and clinical groups using data collection tools. After the pre-test, the patients in the Roy group were trained 6 times in 3 months, twice a month, at home and in the clinic. Nursing interventions were performed using the Roy Adaptation Model in the trainings. At the end of the third month, the post-test data of both groups were collected. During the study, no training or intervention was given to the patients in the clinical group. The nursing education and interventions of this group were carried out by nurses working in the dialysis clinic within the scope of routine practices.

2.3. Evaluation of Data The data were evaluated with the SPSS 23 package program. Percentage, mean and standard deviation values were given for numerical variables, and frequency distributions were given for categorical variables. Chi-square was used to determine the relationship between categorical variables, the independent sample t-test was used to examine the difference between two groups, and the paired-sample t-test was used to examine the changes in the scale averages measured at two different times over time.

2.4. Ethical Principles Permission was obtained from the ethics committee of the University to conduct the study. Consent was obtained from the patients who participated in our study, which was conducted in accordance with the principles of the Declaration of Helsinki. In addition, interventions were applied to the patients in the clinical group at the end of the study, and a training booklet was given.

ELIGIBILITY:
Inclusion Criteria:

* the absence of hearing and visual impairments that would prevent communication
* no diagnosed psychiatric disorder
* literacy
* Turkish proficiency

Exclusion Criteria:

* Not wanting to voluntarily participate in the study.
* Not meeting the inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2016-11-30 (Actual); Study Completion 2017-07-10 (Actual)

PRIMARY OUTCOMES:
Stress | It was used to determine stress levels before starting the study. After 3 months, the interventions were finished and it was used again to measure stress levels.
  Stress was evaluated with the Hemodialysis Stressor Scale

SECONDARY OUTCOMES:
Psychosocial Adjustment | It was used to determine compliance levels before starting the study. After 3 months, the interventions were finished and again used to measure compliance levels.
  Psychosocial Adjustment was evaluated with the Psychosocial Adjustment to Illness-Self-Report Scale

OTHER OUTCOMES:
Self-Care Power | It was used to determine self-care levels before starting the study. After 3 months, the interventions were finished and it was used again to measure self-care levels.
  Self-Care Power was evaluated with the Self-Care Power Scale

CONTACTS AND LOCATIONS:
Overall Officials: Zeynep GÜNGÖRMÜŞ, phD (Associate Professor), Principal Investigator — University of Gaziantep
Locations (1):
- Gaziantep Şahinbey Research and Application Hospital Hemodialysis Unit, Gaziantep, Şehitkamil, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No